CLINICAL TRIAL: NCT01524731
Title: The Effect of Prophylactic Antiemetic Dexamethasone on Plasma Cortisol Levels After Gynecologic Laparotomy
Brief Title: The Effect of Prophylactic Antiemetic Dexamethasone on Plasma Cortisol Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William Li Pi Shan (Other)
Responsible Party: Sponsor-Investigator, William Li Pi Shan, Assistant Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-149-SDR
Record Dates: First submitted 2012-01-24; First posted 2012-02-02 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Sodium Chloride; Saline Solution; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo group
  Interventions: Drug: Saline
- 4 mg dexamethasone (Active Comparator): 4 mg dexamethasone group
  Interventions: Drug: Dexamethasone
- Dexamethasone 8 mg (Active Comparator): Dexamethasone 8 mg group
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Saline — Normal Saline
  Other Names: Normal Saline
  Arms: Placebo
Drug: Dexamethasone — 4 mg
  Other Names: 4 mg dexamethasone
  Arms: 4 mg dexamethasone
Drug: Dexamethasone — 8 mg
  Other Names: 8 mg dexamethasone
  Arms: Dexamethasone 8 mg

SUMMARY:
Dexamethasone is a synthetic corticosteroid that has been proven to be effective and relatively safe for the prophylaxis of the postoperative nausea and vomiting (PONV).

However, little is known about its effect on the hypothalamic-pituitary-adrenal (HPA) axis after surgery. The investigators hypothesize that it will inhibit the normal physiologic HPA surge and reduce cortisol levels post-operatively ia a dose-dependant fashion. To answer this question, the investigators will conduct a randomized, double-blinded placebo-controlled trial with two different doses of dexamethasone in women undergoing elective gynecologic laparotomy.

DETAILED DESCRIPTION:
Hypothesis:

The investigators hypothesize that preoperative administration of intravenous dexamethasone in non-cancer gynecologic laparotomy will decrease postoperative cortisol levels in a dose-dependent fashion.

Objectives:

To compare the post-operative plasma cortisol and glucose level in patients receiving various single doses of dexamethasone versus placebo at the start of gynecologic laparotomy.

To assess the dose-dependent effect of dexamethasone on postoperative pain, nausea and vomiting in this particular context.

To assess the dose-dependent effect of dexamethasone on length of hospital stay.

Methods:

This will be a prospective, randomised, double-blinded trial with two intervention arms and a placebo-control arm conducted at the Royal Victoria Hospital of the McGill University Health Center, Montreal, Canada.

Patients eligible to participate in the study based on inclusion and exclusion criteria will be approached in the preoperative anesthesia clinic (at least one week before the scheduled operation) and some patients will be recruited on the day of surgery hours before in the waiting room by a study personnel who will not be involved in the patient care the day of the surgery. After addressing the patient's questions and concerns, informed consent will be obtained. The patient, the investigators and the anesthesiologist in charge of the patient will be blinded to group allocation until completion of the study.

After patient recruitment, an intravenous line will be placed inside the operating room. Blood will simultaneously be drawn for a baseline plasma cortisol levels. The patients will receive a single IV bolus dose of dexamethasone 4mg, 8mg or an IV normal saline placebo (based on group allocation by randomization) immediately after induction of anesthesia 8. Anesthetic premedication will comprise of 1mg of midazolam. Induction will be performed using 2-3 mg/kg propofol, 2-3 mcg/kg fentanyl, 0.5-1.0 mg/kg rocuronium. Anesthetic maintenance will be performed through an endotracheal tube using desflurane at a minimum of 1 MAC in an equal air/oxygen mixture. Endtidal carbon dioxide tension will be maintained at 40 mmHg using the appropriate ventilator adjustments. Fluid management consists of crystalloid boluses of 20 mg/kg to replace fasting losses, colloid and blood products as necessary according to the surgical losses. Neostigmine and glycopyrrolate reversal will be used if no train of four twitch exists. Ondansetron 4 mg will be given to all patients prior to tracheal extubation.

In the postoperative anesthesia care unit, dimenhydrinate 25-50 mg, prochlorperazine 10 mg will be used should nausea, vomiting, or retching occur. Pain will be controlled by rectal acetaminophen 325mg-1.3 g. Patient controlled analgesia fentanyl will be administered to all patients at a lockout interval of 7 minutes. In the gynaecological ward, dimenhydrinate will be used to control nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 80 years-old scheduled for non-oncologic gynecologic laparotomy, including fibroid myomectomy, hysterectomy and endometrioma resection

Exclusion Criteria:

* Communication barrier rendering informed consent inadequate
* Pregnancy
* Diabetes mellitus
* Chronic or acute renal failure
* Chronic or acute hepatic failure
* History of chronic opioid use
* History of corticosteroid use more than 3 weeks in the last 6 months (inhaled, oral or intravenous)
* History of disorders of the hypothalamus, pituitary gland and/or adrenal glands
* History of depression and/or bipolar disorder
* History of allergy or sensitivity to dexamethasone or any medication used in the standardised anesthetic care
* American Society of Anesthesiologists Physical Status class of 3 and above.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Post operative cortisol level | 24h post-operation
  The primary outcome is the plasma cortisol level at 24h post-operation.

SECONDARY OUTCOMES:
plasma cortisol | 72 hours post-operatively
  Plasma cortisol levels at 6, 48 and 72 hours
Post operative nausea and vomiting scale | 72 hours post-operatively
  Post operative nausea and vomiting at 6, 24, 48 and 72 hours
Post operative pain score | 72 hours post operatively
  postoperative pain scores at 6, 24, 48 and 72 hours
Blood glucose level | 72 hours post-operatively
  blood glucose levels at 6, 24, 48 and 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: William K. Li Pi Shan, MD, Principal Investigator — McGill University
Locations (2):
- Canada (2):
  - McGill University Health Centre-Royal Victoria Hospital, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec